CLINICAL TRIAL: NCT03234062
Title: Developing a Biomarker Panel to Assess Choline Nutritional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 17-0321
Record Dates: First submitted 2017-07-19; First posted 2017-07-31 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Healthy volunteers (n=20), will consume meals, provided by the investigator, in two week intervals with 3 different levels of choline (Cho). Participants will receive 100% of the recommended daily intake (RDI) of Cho (550 mg Cho/day); 50% of the RDI of Cho (275mg/day); and 25% of the RDI of Cho (137.5 mg/day). The meal order will be randomly assigned and all participants will receive all diets at some point in the study. There will be a minimum of a two week washout between diet intervals where participants return to their regular diets. Both participants and researchers will be blinded to the diet order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant dietary arm assignment is randomized by a randomization plan created by the study coordinator at www.randomization.com. Each of the 3 hormonal related demographic groups (male, premenopausal females, and postmenopausal females) will have a list of the same order of diets created by the randomizer. Each participant will be assigned upon entry into the study into the next open diet for their group as ordered by the randomizer. No one collecting or processing data will be informed of the choline levels the participant is experiencing in their dietary arms at any given time to attempt to eliminate bias and ensure appropriate data collection. All staff who interact with participants or who are handling samples/data, will not be informed of the code linking dietary choline levels to diet order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 25%Cho, 50%Cho, 100%Cho (Experimental): Diets containing 137.5mg (25% Cho diet), 275mg (50% Cho diet), and 550mg (100% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 25% Cho, 100% Cho, 50% Cho (Experimental): Diets containing 137.5mg (25% Cho diet) , 550mg (100% Cho diet), and 275mg Cho (50% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 50% Cho, 25% Cho, 100% Cho (Experimental): Diets containing 275mg (50% Cho diet), 137.5mg (25% Cho diet), and 550mg Cho (100% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 50% Cho, 100% Cho, 25% Cho (Experimental): Diets containing 275mg (50% Cho diet), 550mg (100% Cho diet), and 137.5mg Cho (25% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 100% Cho, 25% Cho, 50% Cho (Experimental): Diets containing 550mg (100% Cho diet), 137.5mg (25% Cho diet), and 275mg Cho (50% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet
- 100% Cho, 50% Cho, 25% Cho (Experimental): Diets containing 550mg (100% Cho diet), 275mg (50% Cho diet), and 137.5mg Cho (25% Cho diet) will be given in that order for two weeks each with 2 weeks of washout between.
  Interventions: Other: 25% Cho diet; Other: 50% Cho diet; Other: 100% Cho diet

INTERVENTIONS:
Other: 25% Cho diet — Subjects will consume meals containing 25% of the recommended intake of Choline (137.5 mg Choline/day) for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride-(trimethyl-d9, 9%, Cambridge Isotope Laboratories, Tewksbury, Massachusetts, (USA), as a bolus.
  Other Names: 137.5mg Choline/day
Other: 50% Cho diet — Subjects will consume meals containing 50% of the recommended intake of Choline (275 mg Choline/day) for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride-(trimethyl-d9, 9%, Cambridge Isotope Laboratories, Tewksbury, Massachusetts, (USA), as a bolus.
  Other Names: 275mg Choline/day
Other: 100% Cho diet — Subjects will consume meals containing 100% of the recommended intake of Choline (550 mg Choline/day) for 2 weeks. On day 12 of the diet period, subjects will consume 250 mg of Cho in the form of Cho chloride-(trimethyl-d9, 9%, Cambridge Isotope Laboratories, Tewksbury, Massachusetts, (USA), as a bolus.
  Other Names: 550mg Choline/day

SUMMARY:
People who eat diets low in choline (LC) should deplete their choline (Cho) stores, and measurements of Cho pool size using isotope dilution should reflect this depletion. Investigators will identify a biomarker panel that correlates well with measured Cho pool size across the range of different degrees of depletion.The investigators propose that, as body stores of Cho diminish, cells and organs will reach the point when metabolism/function in the cell is altered, and that this will result in a progression of changes in biomarkers that reflect Cho status.

DETAILED DESCRIPTION:
Choline (Cho) is an essential nutrient and most Americans' diets do not achieve the recommended intake. Diets low in Cho are associated with liver and muscle disease and with suboptimal fetal development, while diets too high in choline may be associated with increased risk for heart disease. Cho is a required nutrient and in 1998, an Adequate Intake (AI) and a Tolerable Upper Limit (UL) for Cho was established In 2016, the US Food and Drug Administration (FDA) set a Recommended Daily Intake (RDI) for Cho based on the AIs as part of the new Nutrition Facts label for packaged foods (published in the Federal Register on May 27, 2016; FDA-2012-N-1210-0875, Federal Register Number:2016-11867). The AI/RDI varies by age and gender, but is 550 mg/d in adolescent and adult men and 425 mg/d in adult women (more in pregnant and lactating women) and 400 mg/day for adolescent women.

There is no validated biomarker for choline status (the availability of the various forms of Cho needed to sustain optimal cellular function). Measurement of plasma Cho concentrations is not adequate as plasma choline is homeostatically regulated. Based on extensive preliminary and published data this group identified a panel of potential biomarkers that could be used to assess Cho status, and now they propose studies to validate this biomarker panel against measures of Cho pool size using isotope dilution. The largest stores of Cho are located in the liver, and mass resonance spectroscopy (MRS) of liver has been used in the past to assess Cho status in humans. This method is not practical for use as a biomarker in clinical or public health practice as it is expensive and the availability of the instrumentation is limited. Liver biopsy is risky and not practical, making measurement of hepatic Cho and Cho metabolites concentrations a poor choice for assessing Cho status.

Perhaps there is a panel of biomarkers that together will more accurately and reliably reflect Cho status. By making measurements in people fed 3 different dietary amounts of Cho for two weeks at a time, and comparing the biomarker measures to body total Cho pool size assessed using isotope dilution (a proxy for the availability of the various forms of Cho), investigators will be able to identify the combination of biomarkers and algorithm for calculating a Cho status score that best predicts total Cho pool size, and therefore predicts choline nutritional status (the availability of the various forms of Cho needed to sustain cellular function). In this pilot study, they are seeking to test a method for using stable isotope dilution to measure body choline stores, and then ask how this measure correlates with a panel of biomarkers in plasma and with liver fat measured using Fibroscan®. Using isotope dilution can provide an estimate of the size of the body pool of Cho. Our proposed method is conceptually similar to the method for measuring total body water from a bolus dose of labeled water. Similar methodology was used recently in studies of metabolic flux of Cho in pregnant women. Isotope dilution is a well-established method used to estimate pool size for other nutrients, such as vitamin A. Similar to vitamin A, the major storage pools for Cho are in the liver, and ingested Cho is rapidly absorbed and accumulated by liver. This pilot study tests a method for using stable isotope dilution to measure body choline stores, and it correlates this measure with a panel of biomarkers in plasma and with liver fat measured using Fibroscan®. People who eat diets low in choline should deplete their choline (Cho) stores, and measurement of Cho pool size using isotope dilution should reflect this depletion. The investigator will identify a biomarker panel that correlates well with measured Cho pool size across the range of different degrees of depletion. MRS/MRI scans will also be performed to investigate correlation between these "gold standard" measures and the other methods described above.

Participants will be consume meals we provide in two week dietary intervals with 3 different levels of choline with 2 week washout periods between those dietary intervals. Participants will receive 100% of the recommended intake (RDI) of Cho (550mg Cho/day); 50% of the RDI of Cho (275mg/day); and 25% of the RDI of Cho (137.5mg/day). The meal order will be randomly assigned and all participants will receive all diets at some point in the study. There will be a minimum of a two week washout between diet intervals. Both participants and researchers will be blinded to the diet order.

Participants will have brief exercise challenges (Biodex) to assess muscle function as an additional predictor of choline status.

To validate our isotope dilution and Fibroscan measures participants will also complete MRI/MRS scans.

Saliva samples, urine, and stool samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 17-70 years
* In good general health as evidenced by medical history, clinical chemistries, physical exam, and BMI≤ 30
* Women who are included in the study and are of pregnancy potential will have a urine pregnancy test at the beginning and end of each dietary intervention arm and must be using birth control during the study.

Exclusion Criteria:

* using drugs or medication known to be damaging to liver or muscle at typically prescribed doses or that have the potential to alter Cho metabolism (e.g., methotrexate);
* history of hepatic, renal, or other chronic systemic disease.
* subjects with liver abnormalities (e.g.cysts) as determined by ultrasound
* current smokers
* consume >2 alcoholic beverages/d or >14/wk
* substance abusers or drug addicted
* eating unusual diet that would interfere with the study
* food allergies, (e.g., soy) or any problems with eating all foods on required study diet
* using Cho-containing dietary supplements
* women who are breastfeeding, pregnant, or plan to become pregnant due to potential risk to fetus/child of low choline diet
* performing intense exercise of more than 1 hour a day or other intense muscle building exercise (such as weightlifting beyond low weight repetitions)
* Actively participating in other research study where required to exercise or ingest any food, medicine, or supplement in any manner
* claustrophobia
* has a cardiac pacemaker, artificial heart valve, metal plate, pin, or other metallic implant, intrauterine device, insulin or other drug pump, aneurysm clips, previous gunshot wound, cochlear implant or other implantable hearing device, employment history as a metalworker, or permanent cosmetic tattoos (eyeliner, eyebrow)

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Change in biomarker panel measures and MRS/MRI scans correlated to different dietary choline levels | Samples taken on Day 12 and Day 14
  The investigator will evaluate direct measures of Choline derived pools and using isotope dilution will provide an estimate of the size of the body pool of choline, while also profiling choline-related metabolites. MRS/MRI will assess Cho compounds in liver and fatty liver (also used to validate Fibroscan) to confirm measures utilizing isotope dilution.

SECONDARY OUTCOMES:
Genotyping for choline metabolism single nucleotide polymorphisms | At baseline visit
  Investigators will ask whether single nucleotide polymorphisms that create inefficiencies in choline metabolism are also associated with decreased choline pool size. SNPs acquired through DNA collection from saliva.
Metabolomic profiling to enhance Cho status score | Samples taken on Day 15
  Untargeted metabolic profiling completed on plasma and urine samples to explore whether there are metabolites detected that enhance Cho status score so that it better predicts Cho pool size as measured using isotope dilution and/or MRS/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Zeisel, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No